CLINICAL TRIAL: NCT06740370
Title: TACE Combined With Lenvatinib and PD-1 Inhibitor for Spontaneous Rupture of Hepatocellular Carcinoma: a Prospective Multicenter Study
Brief Title: TACE Combined With Lenvatinib and PD-1 Inhibitor for Ruptured Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhou Qunfang, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Liver Projiect 14
Record Dates: First submitted 2024-12-13; First posted 2024-12-18 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma; Transcatheter Arterial Chemoembolization; Anti-PD1 Antibody; Lenvatinib
Keywords: ruptured hepatocellular carcinoma; TACE; Lenvatinib; Tislelizumab; Sintilimab; Camrelizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE plus Lenvatinib and PD-1 inhibitor (Experimental): TACE was first performed, then Lenvatinib and PD-1 inhibitor were administered within seven days.
  Interventions: Procedure: TACE; Drug: Lenvatinib; Drug: PD-1 Inhibitors

INTERVENTIONS:
Procedure: TACE — TACE procedure was a 2.8-F microcatheter was super-selectively inserted into the tumor feeding artery using the coaxial technique. Then a combination of lipiodol (5-15 ml), lobaplatin (30-50 mg), and Pirarubicin (30-50 mg) was infused into each tumor. We defined technical success as complete embolization of the tumor-feeding artery resulting in no tumor staining observed by angiogram at the end of procedure.
Drug: Lenvatinib — (12 mg (body weight ≥60 kg) , 8 mg (body weight <60 kg) orally once a day
Drug: PD-1 Inhibitors — Tislelizumab (200mg intravenously every 3 weeks), Sintilimab (200mg intravenously every 3 weeks), Camrelizumab (200mg intravenously every 3 weeks)

SUMMARY:
Hepatocellular carcinoma (HCC) with spontaneous rupture is a potentially fatal complication and usually has poor prognosis. In most conditions, the tumors could not be radically moved. Then minimally therapy like transcatheter arterial chemoembolization (TACE) could effectively stanch the ruptured tumor and bleeding vessels. Then TACE combined the Lenvatinib and PD-1 inhibitor for this subtype HCC could effectively inhibit the tumor and improve the prognosis.

DETAILED DESCRIPTION:
Spontaneous rupture of HCC is a life-threatening complication. HCC rupture is considerably higher in China. The tumor size in ruptured HCC is significantly greater than that in non-ruptured HCC. In the acute phase, hemostasis is the first concern and then tumor treatment is secondary. TACE can effectively induce hemostasis. Conservative treatment is usually system therapy for unresectable ruptured HCC. Thus, we conduct this multicenter single arm study to explore the efficacy, safety of TACE combined lenvatinib and PD-1 inhibitor for unresectable ruptured HCC. This study focuses on the efficacy of TACE combined with lenvatinib and PD-1 inhibitor as first-line therapy.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of primary HCC, confirmed histologically or clinically according to the criteria of the American Association for the Study of Liver Diseases;
2. presence of hemostasis in the enhanced CT scan;
3. integrity of the tumor is disrupted and there is hematoma around the liver;
4. receipt of Lenvatinib and PD-1 inhibitor as the first-line systemic therapy;
5. transarterial artery chemoembolization (TACE) as local therapy;
6. classified as Child-Pugh class A or B and having an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 2;
7. no history of other malignancies.
8. life expectancy more than 3 months;
9. agreed to participated in this clinical trial;
10. Hemameba ≥3.0 x109/L, neutrophil ≥1.5x109/L, hemoglobin≥10.0 g/L, platelet≥100x 109/L, ALT; AST; bilirubin ≤1.5-fold normal, GFR≥60ml/min.

Exclusion Criteria:

1. recurrent HCC;
2. non-ruptured HCC;
3. Lenvatinib and PD-1 inhibitor treated with as second systemic therapy;
4. age < 18 years or > 75 years;
5. HCC with more than five metastases;
6. History of hepatic encephalopathy and gastrointestinal bleeding
7. life expectancy less than 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival (PFS) | 12 months
  Progression was defined as progressive disease by independent radiologic review

SECONDARY OUTCOMES:
Objective response rate (ORR) | 12 months
  ORR, as determined based on tumor response according to mRECIST, is defined as the proportion of all included patients whose best overall response including complete response or partial response.
Overall survival (OS) | 12 months
  OS is the length of time from the date of inclusion until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Duan, MD, Study Director — Chinese PLA General Hospital
Locations (1):
- Qunfang Zhou, Beijing, None Selected, China

IPD SHARING:
Plan to Share IPD: No